CLINICAL TRIAL: NCT03084042
Title: Emotional Brain Networks & Cognitive Functioning in Depression and Anxiety
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Electronic Science and Technology of China (Other)
Collaborators: Sichuan Provincial People's Hospital (Other); The Fourth People's Hospital of Chengdu (Other)
Responsible Party: Principal Investigator, Benjamin Becker, Professor, University of Electronic Science and Technology of China
Other Study IDs: UESTC-neuSCAN-23
Record Dates: First submitted 2017-02-24; First posted 2017-03-20 (Actual); Last update posted 2018-10-29 (Actual); Status verified 2018-10

CONDITIONS: Major Depressive Disorder; General Anxiety Disorder
Keywords: emotional impairments; cognitive impairments
MeSH Terms: conditions — Depressive Disorder, Major; Generalized Anxiety Disorder; Cognitive Dysfunction | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: None Retained — saliva
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Depression patients (MDD): Patients with diagnosis of major depression according to DSM criteria
  Interventions: Device: fMRI
- Anxiety patients (GAD): Patients with generalized anxiety disorder according to DSM criteria
  Interventions: Device: fMRI
- Healthy controls: Demographically matched healthy controls.
  Interventions: Device: fMRI

INTERVENTIONS:
Device: fMRI

SUMMARY:
This study aims to 1) examine common and specific emotional and cognitive dysfunctions between Major Depression and generalized anxiety disorder; 2) Examine emotional and cognitive dysfunctions between the two disorders and healthy controls; 3) Examine the biomarkers predicting successful therapy or not.

ELIGIBILITY:
Inclusion Criteria:

* GAD:

  1. Diagnosis of Generalized Anxiety Disorder (GAD) according to DSM V criteria in a structured clinical interview for DSM-V Axis I disorders (SCID I; APA, 2014) and a confirmatory clinical interview
  2. Duration of the current episode > 3 weeks
* MDD:

  1. Diagnosis of current major depressive disorder in a structured clinical interview for DSM-V Axis I disorders (SCID I; APA, 2014) and a confirmatory clinical interview
  2. Duration of the current episode > 4 weeks

Exclusion Criteria:

* GAD: diagnosis of any other psychiatric Axis I disorder (except GAD) as a principal diagnosis within the past six months
* MDD: diagnosis of any other psychiatric Axis I disorder (except MDD) as a principal diagnosis within the past six months

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients from the hospitals and healthy controls from community
Sampling Method: Non-Probability Sample
Enrollment: 105 (Estimated)
Dates: Start 2016-07; Primary Completion 2018-12 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Brain activity in the emotional and cognitive core regions of the brain as assessed by fMRI | 1 hour (assessed at study inclusion)
  fMRI based indices during emotional face processing
Brain activity in the emotional and cognitive core regions of the brain as assessed by fMRI | 1 hour (assessed at study inclusion)
  fMRI based indices during empathy processing
Brain activity in the emotional and cognitive core regions of the brain as assessed by fMRI | 1 hour (assessed at study inclusion)
  fMRI based indices during working memory

SECONDARY OUTCOMES:
Behavioral performance during the fMRI: face processing | 1 hour (assessed at study inclusion)
  Accuracy during face processing
Behavioral performance during the fMRI: empathy reactivity | 1 hour (assessed at study inclusion)
  Empathy in response to empathy inducing pictures (rated on Likert scale)
Behavioral performance during the fMRI: working memory | 1 hour (assessed at study inclusion)
  Working memory performance during fMRI
Cognitive performance at study inclusion | 1 hour (assessed at study inclusion)
  Executive functions as assessed via computerized tests (CANTAB)
Symptom improvement after 3 months: depression | 3 months
  Symptoms of depression will be assessed using validated clinical scales (e.g. BDI)
Symptom improvement after 3 months: anxiety | 3 months
  Symptoms of generalized anxiety will be assessed using validated clinical scales (e.g. Penn State Worry Questionnaire)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Becker, Dr., Principal Investigator — School of Life Science and Technology, University of Electronic Science and Technology of China
Locations (1):
- School of Life Science and Technology, University of Electronic Science and Technology of China, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No